CLINICAL TRIAL: NCT02636478
Title: Travel Activities in Patients With Sleep Related Breathing Disorders
Brief Title: Travelling in Patients With Sleep Related Breathing Disorders
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Responsible Party: Sponsor
Other Study IDs: WI_23/2013
Record Dates: First submitted 2015-11-02; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Travel, Sleep Related Disorder
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- reference group: therapy naive patients with a sleep related breathing disorder
  Interventions: Other: questionnaire for travel habits
- therapy group: patients with devices treating their sleep related breathing disorder
  Interventions: Other: questionnaire for travel habits

INTERVENTIONS:
Other: questionnaire for travel habits — questionnaire has been used to collect information about travelling

SUMMARY:
One questionnaire has been configured to ask therapy naive and treated patients about their travel activities. Travel activities include private and professional traveling. Another questionnaire collects medical information.

DETAILED DESCRIPTION:
Including a German sleep committee a new questionnaire has been created to ask patients about their travel Habits. Only travels over a onenightstay were of interest. All detailed Information about the Destination has been asked. A Special Point of interest were the Impacts of traveling. For each Patient a doctor completed the medical history including sleep related breathing disorder and relevant medical conditions e.g. orthopedic Impacts.

ELIGIBILITY:
Inclusion Criteria:

* patients with sleep related breathing disorder
* informed consent provided

Exclusion Criteria:

* patients with no sleep related breathing disorder
* no informed consent provided

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with sleep related breathing disorder
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
travel activities in sleep related breathing disorder, questionnaire | ten minutes
  questionnaire has been used once in each patient

REFERENCES:
- [Background] Quera Salva MA, Barbot F, Hartley S, Sauvagnac R, Vaugier I, Lofaso F, Philip P. Sleep disorders, sleepiness, and near-miss accidents among long-distance highway drivers in the summertime. Sleep Med. 2014 Jan;15(1):23-6. doi: 10.1016/j.sleep.2013.06.018. Epub 2013 Sep 14. PMID 24286897
- [Background] Sinagawa DM, De Carvalho HB, Andreuccetti G, Do Prado NV, De Oliveira KC, Yonamine M, Munoz DR, Gjerde H, Leyton V. Association between travel length and drug use among Brazilian truck drivers. Traffic Inj Prev. 2015;16(1):5-9. doi: 10.1080/15389588.2014.906589. Epub 2014 Sep 26. PMID 24697351